CLINICAL TRIAL: NCT02186730
Title: Computerised Intervention/Treatment for Adolescent Depression and Low Mood: Feasibility Phase 2
Brief Title: Computerised Intervention/Treatment for Adolescent Depression and Low Mood:
Acronym: CITADAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leeds and York Partnership NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CITADAL
Record Dates: First submitted 2014-06-25; First posted 2014-07-10 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Depression
Keywords: Computerised Cognitive Behaviour Therapy; Adolescents; Depression; Low Mood
MeSH Terms: conditions — Depression; Consciousness Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stressbsuters (Experimental): Computerised Cognitive Behaviour package consisting of eight 30-45 minute sessions of CBT designed for 12-18 year olds. Each Stressbusters session is an interactive presentation featuring narration synchronised with videos, animations, graphics and printouts.
  The programme has a narrator guiding individuals through each of the eight sessions in a linear progression. Each session builds on the knowledge gained in previous sessions and on tasks carried out at home. Sessions contain flexible "add-ons" such as written fact sheets (for example about bullying, sleep problems) which can be printed out and taken away together with home practice related handouts from the programme (for example mood diary sheets). Session topics include getting activated, relapse prevention, challenging negative thoughts and problem solving
  Interventions: Behavioral: Stressbusters
- Websites (Active Comparator): Any individuals randomised to arm 2 of the trial will spend the equivalent time accessing currently available self help websites that provide information about low mood/depression. These four websites will be the same as those used in our initial feasibility study of which, based on our preliminary data, there is evidence for their usefulness.
  Interventions: Behavioral: Websites

INTERVENTIONS:
Behavioral: Stressbusters — cCBT
  Arms: Stressbsuters
Behavioral: Websites — Self help websites
  Arms: Websites

SUMMARY:
This study forms the second phase of previous work to examine the effectiveness of computerised Cognitive Behaviour Therapy (cCBT) to treat adolescents with low mood/depression.

Depression affects around 2% of adolescents. Antidepressants are not recommended for this age range as a first line treatment because of concerns about their usefulness and side effects. Government guidelines have supported using Cognitive Behaviour Therapy (CBT), which is effective and one of the main treatments recommended for depression. It has been suggested that computerised versions of CBT (cCBT) may be effective for treating depression in young people who may prefer this to seeing a therapist face-to-face, but little research exists to date to support this. This study examines the feasibility of running a large scale randomised controlled trial (RCT) to compare a promising cCBT program (Stressbusters) with self-help websites for adolescents with low mood and depression (LMD).

Eligible and consenting participants will complete several questionnaires to assess their mood before being randomly assigned to either cCBT (Stressbusters) or equivalent access to selected websites providing self help for LMD. Participants will complete further mood questionnaires 4 and 12 months after treatment completion/withdrawal. We have already recruited 97 individuals to this trial but aim to recruit a further 48 participants to collect further information.

We are also keen to find out whether sending participants text messages before sessions and around follow up periods will increase attendance/completion. Therefore all trial participants will receive text messages from the research team during their participation.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 18 years
* Low mood/depression
* co-morbid physical illness or co-morbid non-psychotic functional disorders, such as anxiety

Exclusion Criteria:

* Suicidality
* Postnatally depressed
* Suffering psychotic symptoms

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2014-04-03 (Actual); Primary Completion 2015-04-27 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
Changes on the Short Beck Depression Inventory from baseline to 4 and 12 months follow up | baseline, 4 months follow up, 12 months follow up

SECONDARY OUTCOMES:
Changes on the Mood and Feelings Questionnaire from baseline to 4 and 12 months follow up | Baseline, 4 months follow up, 12 months follow up
The Short Mood and Feelings Questionnaire | up to 8 weeks
Changes on the Spence Children's Anxiety Scale from baseline to 4 and 12 months follow up | Baseline, 4 months follow up and 12 months follow up
Changes in health status measured by the EQ-5D-Y from baseline to 4 and 12 months follow up | Baseline, 4 months follow up, 12 months follow up
Changes in health status measured by the HUI2 from baseline to 4 and 12 months follow up | Baseline, 4 months follow up and 12 months follow up
The number of health services used by participants between baseline, 4 months and 12 months follow up | Baseline, 4 months follow up, 12 months follow up

OTHER OUTCOMES:
Further mental health support received during trial participation | 12 months
Number of self-harm episodes during trial participation | 12 months
Number of inpatient admissions during trial participation | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Barry Wright, Principal Investigator — LYPFT
Locations (1):
- Limetrees Child Adolescent and Family Unit, York, North Yorkshire, United Kingdom